CLINICAL TRIAL: NCT00532922
Title: A 3-Month Non-Interventional Study of Asthmatics Treatment With Symbicort® Turbuhaler®
Acronym: Symb NIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-RCN-SYM-2006/1
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Chinese asthma patient prescribed Symbicort® Turbuhaler®

SUMMARY:
The purpose of this study is to investigate real practices of treatment with Symbicort Turbuhaler for 3 months in asthma and patient compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Asthmatics who has been prescribed Symbicort according to physician's judgement
3. Usage of Symbicort should follow local prescribing information

Exclusion Criteria:

1. Not being involved in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site)
2. No previous enrolment in the present study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Natural History, longitudinal, defined population
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2007-04; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Xin, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Hong Jianguo, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (19):
- China (19):
  - Research Site, Hefel, Anhui
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Wuhan, Hubel
  - Research Site, Nanjong, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Shenyand, Liaoning
  - Research Site, Qingdao, Shandong
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Wenzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Hangzhou
  - Research Site, Shanghai